CLINICAL TRIAL: NCT05580146
Title: Acute Dose-ranging Effects of Mango Leaf Extract (Zynamite® 15%) on Cognitive Function and Cerebral Blood Flow in Healthy Young Adults
Brief Title: Acute Dose-ranging Effects of Mango Leaf Extract (Zynamite® 15%) on Cognitive Function and Cerebral Blood Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Nektium Pharma SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 58BX2 and 58BX3
Record Dates: First submitted 2021-05-05; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-04

CONDITIONS: Cognitive Change
Keywords: NIRS; Cognitive Performance; Cerebral Blood Flow; Mango Leaf Extract; Zynamite®; Mangifera indica
MeSH Terms: interventions — Mangifera indica extract

STUDY DESIGN:
Intervention Model Description: Balanced crossover
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Zynamite® 15% 150mg (Active Comparator): Mango leaf extract (Mangifera indica)
  Interventions: Dietary Supplement: Zynamite® 15% 150mg
- Zynamite® 15% 300mg (Active Comparator): Mango leaf extract (Mangifera indica)
  Interventions: Dietary Supplement: Zynamite® 15% 300mg
- Zynamite® 15% 600mg (Active Comparator): Mango leaf extract (Mangifera indica)
  Interventions: Dietary Supplement: Zynamite® 15% 600mg
- Placebo (Placebo Comparator): Placebo matched for appearance
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Zynamite® 15% 150mg — leaves of the mango food plant
  Other Names: Mangifera indica
  Arms: Zynamite® 15% 150mg
Dietary Supplement: Zynamite® 15% 300mg — leaves of the mango food plant
  Other Names: Mangifera indica
  Arms: Zynamite® 15% 300mg
Dietary Supplement: Zynamite® 15% 600mg — leaves of the mango food plant
  Other Names: Mangifera indica
  Arms: Zynamite® 15% 600mg
Dietary Supplement: Placebo — Sunflower oil matched for appearance
  Arms: Placebo

SUMMARY:
Zynamite® is a novel mango (Mangifera indica) leaf extract standardized to contain polyphenol mangiferin.It has previously been shown to enhance brain oxygenation, physical performance and ergogenic parameters following ischemia-reperfusion in healthy humans when consumed alongside other polyphenols. Preliminary data has also indicated that a single 300mg dose of Zynamite® (60%) can improve performance across a range of cognitive tasks.This study aims to evaluate the effects, in healthy adults, of 3 doses of Zynamite® 15% on performance across a number of cognitive domains, as well as during a period of cognitively demanding task performance. A second sub-study will assess cerebral blood flow during cognitively demanding task performance.

DETAILED DESCRIPTION:
Extracts made from the leaves of the mango food plant (Mangifera indica L., Anacardiaceae) have a long history of medicinal usage, most likely due to particularly high levels of the polyphenol mangiferin. Zynamite®, is a novel mango (Mangifera indica) leaf extract standardized to contain polyphenol mangiferin which has previously been shown to enhance brain oxygenation and physical performance and ergogenic parameters following ischemia-reperfusion in healthy humans when consumed alongside other polyphenols.A recent study in rats demonstrated a similar effect of Zynamite® on electrophysiological (EEG) spectral power as that seen following caffeine, with a synergistic effect of co-consumption of Zynamite® and caffeine. A concomitant ex vivo study demonstrated increased long-term potentiation (LTP) in rat hippocampal slices, suggesting the potential for Zynamite® to enhance memory. Previous research has also demonstrated that both single doses and chronic administration of polyphenols can beneficially modulate cognitive function, including during cognitively demanding task performance. Previous research has also shown that polyphenols and polyphenol rich treatments can modulate cerebral blood-flow. These findings raise the possibility that Zynamite® may have beneficial effects on psychological and hemodynamic parameters, potentially with some similarities to the effects exerted by caffeine.

A recent study expanded on the above assessing the effects of a single dose of Zynamite® (60% of polyphenol mangiferin) on performance across a number of cognitive domains (attention, working memory, episodic memory, executive function), as well as during a period of cognitively demanding task performance, and during laboratory-induced stress. The results showed that a single dose of 300 mg Zynamite® significantly improved performance accuracy across the tasks in the battery, with domain-specific effects seen in terms of enhanced performance on an 'Accuracy of Attention' factor and an 'Episodic Memory' factor as well as improved performance across all three tasks (Rapid Visual Information Processing, Serial 3s and Serial 7s subtraction tasks) of the Cognitive Demand Battery sub-section of the assessment, which assesses cognitive function and subjective mental fatigue during sustained performance of mentally demanding tasks. All of these cognitive benefits were seen across the post-dose assessments (30 min, 3 h, 5 h). These results provide the first demonstration of cognition enhancement following consumption of mango leaf extract adding to previous research showing that polyphenols and polyphenol rich extracts can improve brain function.

The proposed studies will expand on the existing body of research by assessing the effects of three doses of Zynamite® (this time a lower concentration version containing 15% polyphenol mangiferin) on cognitive performance and cerebral blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Participants must self-assess themselves as being in good health
* Participants must be aged 18 to 30 years at the time of giving consent
* Participants must self-report playing video-games (arcade, console, computer, smartphone) for not less than 5 hours a week on average, over the previous 6 months .

Exclusion Criteria:

* Have symptoms of Covid-19 or fall into the 'high' or 'moderate' risk categories from coronavirus as defined by NHS UK.
* Have any pre-existing diagnosed medical condition/illness which will impact taking part in the study NOTE: the explicit exception to this is controlled hay fever. There may be other, unforeseen, exceptions and these will be considered on a case-by-case basis; i.e. participants may be allowed to progress to screening if they have a condition/illness which would not interact with the active treatments or impede performance. Note asthma is not permitted in this study.
* Are currently taking prescription medications including habitual use of non-steroidal anti-inflammatory drugs (NSAIDs) (e.g. ibuprofen, aspirin) NOTE: the explicit exceptions to this are contraceptive treatments for female participants, thyroid medication, topical creams and those taken 'as needed' in the treatment of hay fever. As above, there may be other instances of medication use which, where no interaction with the active treatments is likely, and which would not be expected to have any impact on brain function, participants may be able to progress to screening.
* Have high blood pressure (systolic over 139 mm Hg or diastolic over 89 mm Hg)
* Have a Body Mass Index (BMI) outside of the range 18.5-29.9 kg/m2
* Are pregnant, seeking to become pregnant or lactating.
* Have learning and/or behavioural difficulties such as dyslexia or ADHD
* Have a visual impairment that cannot be corrected with glasses or contact lenses (including colour-blindness)
* Smoke tobacco or vape nicotine or use nicotine replacement products
* Excessive caffeine intake (>500 mg per day)
* Have relevant food intolerances/ sensitivities/ allergies
* Have taken antibiotics within the past 4 weeks
* Have taken dietary supplements e.g. vitamins, omega 3 fish oils etc. in the last 4 weeks (Note: participation is possible following a 4 week supplement washout prior to participating and for the duration of the study on the proviso that the supplements they are taking are out of choice and not medically prescribed or advised). NOTE: Existing vitamin D use is permitted
* Have any health condition that would prevent fulfilment of the study requirements (this includes non-diagnosed conditions for which no medication may be taken)
* Are unable to complete all of the study assessments
* Are currently participating in other clinical or nutrition intervention studies, or have in the past 4 weeks
* Has been diagnosed with/ undergoing treatment for alcohol or drug abuse in the last 12 months
* Have been diagnosed with/ undergoing treatment for a psychiatric disorder in the last 12 months
* Suffers from frequent migraines that require medication (more than or equal to 1 per month)
* Sleep disorders or are taking sleep aid medication
* Any known active infections
* Does not have a bank account (required for payment)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
Cerebral blood flow during performance of cognitive tasks | 60 minutes post-dose
  Measured (in umol) using quantitative near infrared spectroscopy (higher indicates increased blood volume)
Cerebral blood flow at rest | 10 minutes
  Measured (in umol) using quantitative near infrared spectroscopy (higher indicates increased blood volume)
Change in speed of performance from baseline to 300 minutes post dose | 0, 300 minutes post dose
  This is a composite measure derived from summing the z score reaction time (RT) performance on seven tasks and finding the average: Speed of performance = (Zsimple RT + Zchoice RT + Zdigit vigilance RT + ZRVIP RT + ZNumeric working memory RT + ZPicture recognition RT + ZWord recognition RT) ÷ 7
Change in accuracy of cognitive task performance from baseline to 300 minutes post dose | 0, 300 minutes post dose
  This is a composite measure derived from summing the z score accuracy performance scores on nine tasks and finding the average: Accuracy of performance = (Zaccuracy choice RT + Zdigit vigilance accuracy + ZRVIP accuracy + ZNumeric working memory accuracy + ZCorsi span score + Zimmediate word recall accuracy + Zdelayed word recall accuracy + Zword recognition accuracy + Zpicture recognition accuracy) ÷ 9
Change in accuracy of attention from baseline to 300 minutes post dose | 0, 300 minutes post dose
  This is a composite measure derived from averaging the sum of the the z score accuracy performance scores from the choice reaction time, digit vigilance and Rapid visual information processing tasks
Change in speed of attention from baseline to 300 minutes post dose | 0, 300 minutes post dose
  This is a composite measure derived from averaging the sum of the the z score reaction times from the choice reaction time, digit vigilance and Rapid visual information processing tasks
Change in working memory from baseline to 300 minutes post dose | 0, 300 minutes post dose
  This is a composite measure derived from averaging the sum of the z score accuracy performance on the numeric working memory task and Corsi block-tapping task
Change in speed of memory from baseline to 300 minutes post dose | 0, 300 minutes post dose
  This is a composite measure derived from averaging the sum of the z score reaction times on the numeric working memory task, the delayed picture recognition task and the delayed word recognition task
Change in episodic memory from baseline to 300 minutes post dose | 0, 300 minutes post dose
  This is a composite measure derived from averaging the sum of the z score performance on the following cognitive tasks: immediate word recall, delayed word recall, delayed picture recognition, delayed word recognition
Cognitive function- change in individual task Accuracy for word recall from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Task Accuracy
Cognitive function- change in individual task Accuracy for word recognition from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Task Accuracy
Cognitive function- change in individual task Accuracy for picture recognition from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Task Accuracy
Cognitive function- change in individual task Accuracy for numeric working memory from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Task Accuracy
Cognitive function- change in individual task Accuracy for choice reaction time from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Task Accuracy
Cognitive function- change in individual task Accuracy for digit vigilance from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Task Accuracy
Cognitive function- change in individual task Accuracy for corsi blocks task from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Task Accuracy
Cognitive function- change in individual task Accuracy for peg and ball from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Task Accuracy
Cognitive function- change in individual task Reaction Time for picture recognition from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Reaction Time
Change in Reaction Time for word recognition from baseline to 300 minutes post dose Cognitive function- individual task Reaction Time for word recognition Cognitive function- individual task Reaction Time for word recognition | 0, 300 minutes post dose
  Reaction Time
Cognitive function- change in individual task Reaction Time for numeric working memory from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Reaction Time
Cognitive function- change in individual task Reaction Time for choice reaction time from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Reaction Time
Cognitive function- change in individual task Reaction Time for digit vigilance from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Reaction Time
Cognitive function- change in individual task Reaction Time for simple reaction time from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Reaction Time
Cognitive function- change in individual task Reaction Time for peg and ball from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Reaction Time
Cognitive Function- change in serial 3 subtractions accuracy from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Task accuracy
Cognitive Function- change in serial 7 subtractions accuracy from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Task accuracy
Cognitive Function- change in Rapid Information Visual Processing accuracy from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Task accuracy
Cognitive Function- change in Rapid Information Visual Processing reaction time from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Reaction time
Cognitive Function- change in Rapid Information Visual Processing false alarms from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Number of false alarms
Mental fatigue- change in subjective mental fatigue from baseline to 300 minutes post dose | 0, 300 minutes post dose
  Mental fatigue visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: David Kennedy, Prof, Principal Investigator — Northumbria University
Locations (1):
- Brain performance and nutrition research centre, Northumbria university, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No